CLINICAL TRIAL: NCT03364595
Title: Operative Plate Fixation Versus Replacement for Mason Type III Fracture of Radial Head
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Yichong, Department of orthopaedics and trauma, Peking University People's Hospital
Other Study IDs: CSGK-RGXT
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Radial Head Fracture
Keywords: radial head fracture; replacement; plate
MeSH Terms: conditions — Radial Head and Neck Fractures | interventions — Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Plate Fixation: The operating surgeon will determine the positioning of the patient for surgery. ORIF of the radial head fracture will be carried out
  Interventions: Procedure: plate fixation
- Replacement: The operating surgeon will determine the positioning of the patient for surgery. During the surgery, they take out the the comminuted radial head and proceed replacement using artificial.
  Interventions: Procedure: replacement

INTERVENTIONS:
Procedure: plate fixation — ORIF of the radial head fracture
  Groups: Plate Fixation
Procedure: replacement — replacement of the radial head fracture
  Groups: Replacement

SUMMARY:
To compare the effect of Operative Plate Fixation Versus Replacement for Mason Type III Fracture of Radial Head

DETAILED DESCRIPTION:
From April 2015 to October 2016, patients with comminuted radial head fractures diagnosed as Mason type III are retrospectively included in this study, they were treated with either operative plate or radial head replacement. All the patients are regularly followed up in clinic. Then we will compare the union rate and clinical functional outcome(Mayo score) between the 2 groups at 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

Men or women aged 18 to 65 years of age with Mason Type III radial head fracture are confirmed by radiograph within 1 month post injury Provision of informed consent

Exclusion Criteria:

Pathological fractures Non-displaced (cortical contact) fractures Open fractures Presence of vascular or nerve injury Fractures more than 1 month post-injury Limited life expectancy due to significant medical co-morbidity Medical contraindication to surgery Inability to comply with rehabilitation or form completion Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men or women aged 18 to 65 years of age with Mason Type III radial head fracture
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Union rate | 1 year after surgery
  Union rate of the fracture from X-ray

SECONDARY OUTCOMES:
Functional score | 1 year after surgery
  Mayo score of injury elbow

CONTACTS AND LOCATIONS:
Overall Officials: Peixun Zhang, MD, Study Director — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No